CLINICAL TRIAL: NCT02217904
Title: A Single-Dose Clinical Trial to Study the Safety, Tolerability, Pharmacokinetics, and Anti-Retroviral Activity of MK-8591 Monotherapy in Anti-Retroviral Therapy (ART)-Naive, HIV-1 Infected Patients
Brief Title: A Study of Islatravir (MK-8591) in Anti-Retroviral Therapy-Naive, Human Immunodeficiency Virus-1 Infected Participants (MK-8591-003)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8591-003; 2014-002192-28 (EudraCT Number); MK-8591-003 (Other: Merck Protocol Number)
Record Dates: First submitted 2014-08-13; First posted 2014-08-15 (Estimated); Results first posted 2018-12-03 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-07

CONDITIONS: HIV-1
MeSH Terms: interventions — islatravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Islatravir 1 mg (Experimental): Single oral dose of islatravir 1 mg
  Interventions: Drug: 1 mg islatravir
- Islatravir 2 mg (Experimental): Single oral dose of islatravir 2 mg
  Interventions: Drug: 2 mg islatravir
- Islatravir 10 mg (Experimental): Single oral dose of islatravir 10 mg
  Interventions: Drug: 10 mg islatravir
- Islatravir 30 mg (Experimental): Single oral dose of islatravir 30 mg
  Interventions: Drug: 30 mg islatravir
- Islatravir 0.5 mg (Experimental): Single oral dose of islatravir 0.5 mg
  Interventions: Drug: 0.5 mg islatravir
- Islatravir 0.25 mg (Experimental): Single oral dose of islatravir 0.25 mg
  Interventions: Drug: 0.25 mg islatravir
- Islatravir 30 mg Extended Observation (Experimental): Single oral dose of 30 mg islatravir administered following >8 hour fast. Participants will be closely monitored for viral load for up to approximately 21 days prior to starting standard of care ART.
  Interventions: Drug: 30 mg islatravir

INTERVENTIONS:
Drug: 1 mg islatravir — Single oral dose of 1 mg islatravir administered following ≥8 hour fast
  Other Names: MK-8591
  Arms: Islatravir 1 mg
Drug: 2 mg islatravir — Single oral dose of 2 mg islatravir administered following ≥8 hour fast
  Other Names: MK-8591
  Arms: Islatravir 2 mg
Drug: 10 mg islatravir — Single oral dose of 10 mg islatravir administered following ≥8 hour fast
  Other Names: MK-8591
  Arms: Islatravir 10 mg
Drug: 30 mg islatravir — Single oral dose of 30 mg islatravir administered following ≥8 hour fast
  Other Names: MK-8591
  Arms: Islatravir 30 mg; Islatravir 30 mg Extended Observation
Drug: 0.5 mg islatravir — Single oral dose of 0.5 mg islatravir administered following ≥8 hour fast
  Other Names: MK-8591
  Arms: Islatravir 0.5 mg
Drug: 0.25 mg islatravir — Single oral dose of 0.25 mg islatravir administered following ≥8 hour fast
  Other Names: MK-8591
  Arms: Islatravir 0.25 mg

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics, and anti-retroviral therapy (ART) activity of islatravir (MK-8591) monotherapy in ART-naive, human immunodeficiency virus-1 (HIV-1) infected participants. The primary hypothesis is that at a safe and tolerable dose of islatravir, the true mean difference in the plasma HIV-1 ribonucleic acid (RNA) reduction from baseline between islatravir and placebo is at least 0.5 log (base10) copies/mL.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant, non-breast feeding, postmenopausal or surgically sterile female
* Female with reproductive potential agrees to use (or have male partner use) two acceptable methods of birth control
* Male agrees to use acceptable method of contraception during study and for 90 days after last dose of trial drug
* Has stable baseline health, other than HIV infection
* Has no significantly abnormal electrocardiogram
* Is HIV-1 positive
* Have a screening plasma HIV-1 RNA ≥ 10,000 copies/mL within 30 days prior to the treatment phase of this study. For inclusion in Panel Islatravir Extended Observation, participants must also have a screening plasma HIV-1 RNA ≤ 25,000 copies/mL within 30 days prior to the treatment phase.
* Is ART naive
* Has not received any investigational agent or marketed ART within 30 days of trial drug administration
* Is diagnosed with HIV-1 infection >= 3 months prior to screening
* Is willing to receive no other ART during treatment phase of study
* Has no evidence of mutations conferring resistance to nucleoside reverse transcriptase inhibitors (NRTIs)

Exclusion Criteria:

* Is mentally or legally institutionalized/incapacitated, or has significant emotional problems, or has a history of clinically significant psychiatric disorder of the last 5 years
* Has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological (outside of HIV-1 infection), renal, respiratory, genitourinary, major neurological abnormalities or diseases
* Has a history of cancer (malignancy)
* Has a history of significant multiple and/or severe allergies, or had an anaphylactic reaction to drugs or food
* Is positive for hepatitis B surface antigen
* Has a history of chronic Hepatitis C
* Had major surgery or lost 500 mL of blood with 4 weeks prior to screening visit
* Has participated in another investigational trial within 4 weeks prior to dosing visit
* Will use any medications, prescribed drugs, or herbal remedies 4 weeks prior to dosing of trial drug, up to the post-trial visit
* Consumes excessive amounts of alcohol, caffeinated beverages, or tobacco products
* Uses illicit drugs or has a history of drug abuse within the prior 2 years

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09-17 (Actual); Primary Completion 2017-05-11 (Actual); Study Completion 2017-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Schurmann D, Rudd DJ, Zhang S, De Lepeleire I, Robberechts M, Friedman E, Keicher C, Huser A, Hofmann J, Grobler JA, Stoch SA, Iwamoto M, Matthews RP. Safety, pharmacokinetics, and antiretroviral activity of islatravir (ISL, MK-8591), a novel nucleoside reverse transcriptase translocation inhibitor, following single-dose administration to treatment-naive adults infected with HIV-1: an open-label, phase 1b, consecutive-panel trial. Lancet HIV. 2020 Mar;7(3):e164-e172. doi: 10.1016/S2352-3018(19)30372-8. Epub 2020 Jan 3. PMID 31911147

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Additional panels (F: 0.25 mg islatravir; and G: 30 mg islatravir Extended Observation) were initially planned but were not conducted.
Groups:
- Panel A: 10 mg Islatravir: Participants received a single dose of 10 mg islatravir.
- Panel B: 2 mg Islatravir: Participants received a single dose of 2 mg islatravir.
- Panel C: 30 mg Islatravir: Participants received a single dose of 30 mg islatravir.
- Panel D: 1 mg Islatravir: Participants received a single dose of 1 mg islatravir.
- Panel E: 0.5 mg Islatravir: Participants received a single dose of 0.5 mg islatravir.
- Panel F: 0.25 mg Islatravir: Participants received a single does of 0.25 mg islatravir.
- Panel G: 30 mg Islatravir Extended Observation: Participants received a single does of 30 mg islatravir.
Period: Overall Study
Arm/Group | Panel A: 10 mg Islatravir | Panel B: 2 mg Islatravir | Panel C: 30 mg Islatravir | Panel D: 1 mg Islatravir | Panel E: 0.5 mg Islatravir | Panel F: 0.25 mg Islatravir | Panel G: 30 mg Islatravir Extended Observation
Started | 6 | 6 | 6 | 6 | 6 | 0 | 0
Completed | 6 | 6 | 6 | 6 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Panel A: 10 mg Islatravir | Panel B: 2 mg Islatravir | Panel C: 30 mg Islatravir | Panel D: 1 mg Islatravir | Panel E: 0.5 mg Islatravir | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.5 (10.0) | 42.2 (9.8) | 35.5 (9.1) | 32.7 (12.7) | 35.5 (11.3) | 35.5 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 6 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 1 | 0 | 3
  Not Hispanic or Latino | 4 | 6 | 6 | 5 | 6 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 6 | 6 | 6 | 5 | 6 | 29
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Plasma HIV-1 Ribonucleic Acid (RNA) [Mean (Standard Deviation); unit: log10 copies/mL] | 4.68 (0.39) | 4.7 (0.25) | 4.17 (0.41) | 4.66 (0.2) | 4.59 (0.5) | 4.56 (0.40)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Plasma HIV-1 RNA at 168 Hours Post-Dose
Description: Plasma HIV-1 RNA was measured using the Roche COBAS Ampliprep/COBAS TaqMan HIV-1 test v.2.0, which has a linear range from 20 to 10,000,000 copies/mL. The lower limit of detection has 100% specificity at 20 copies/mL. Additionally, the test increases the probability of detection and expands coverage by targeting two highly conserved regions of the HIV-1 genome to compensate for the possibility of mutations or mismatches.
Time Frame: Baseline and 168 hours (7 days) post-dose
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment, were compliant with study procedures, had available plasma HIV-1 RNA data at baseline and 168 hours post-dose, and were evaluable for the outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 copies/mL
Arm/Group | Panel A: 10 mg Islatravir | Panel B: 2 mg Islatravir | Panel C: 30 mg Islatravir | Panel D: 1 mg Islatravir | Panel E: 0.5 mg Islatravir
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
log10 copies/mL | -1.67 [-1.92 to -1.42] | -1.35 [-1.60 to -1.10] | -1.60 [-1.85 to -1.34] | -1.30 [-1.55 to -1.05] | -1.20 [-1.46 to -0.95]
Statistical Analysis 1: Comparison: Panel A: 10 mg Islatravir; Adjusted by Placebo data pooled from historical placebo data from recent monotherapy studies in HIV-1 infected participants (NCT00100048, NCT01466985, NCT01152255, and NCT01353898) and fitted with a longitudinal data analysis (LDA) model containing fixed effects for study and time, and a random effect for participants. LS mean of pooled historical placebo data was -0.03 log10 copies/mL (95% CI -014, 0.09) change from baseline at 168 hours post dose; Test type: Superiority; Posterior mean difference = -1.64 — Posterior Probability (PP) of true mean difference in the plasma HIV-1 RNA change from baseline between islatravir and placebo at least 0.5 log10 copies/mL was >99%
Statistical Analysis 2: Comparison: Panel B: 2 mg Islatravir; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Posterior mean difference = -1.32 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Panel C: 30 mg Islatravir; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Posterior mean difference = -1.57 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Panel D: 1 mg Islatravir; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Posterior mean difference = -1.28 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Panel E: 0.5 mg Islatravir; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Posterior mean difference = -1.18 — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Number of Participants With One or More Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a study participant administered a pharmaceutical product that does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
Time Frame: Up to 21 days post-dose
Population: All participants who received at least one dose of investigational drug
Measure: Count of Participants; unit: Participants
Arm/Group | Panel A: 10 mg Islatravir | Panel B: 2 mg Islatravir | Panel C: 30 mg Islatravir | Panel D: 1 mg Islatravir | Panel E: 0.5 mg Islatravir
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Participants | 5 | 5 | 6 | 5 | 6

3. Secondary Outcome: Area Under the Concentration-Time Curve of Islatravir Triphosphate in Peripheral Blood Mononuclear Cells From Time 0 to 168 Hours (AUC0-168hr)
Description: Blood was collected to measure intracellular islatravir triphosphate concentration in peripheral blood mononuclear cells and determine AUC0-168hr.
Time Frame: 4, 12, 24, 96, 120, 144, and 168 hours after islatravir administration. Value at predose was inferred from plasma predose sample.
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment, were compliant with study procedures, had AUC0-168hr of triphosphate in peripheral blood mononuclear cells data available, and were evaluable for the outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*pmol/10^6 cells
Arm/Group | Panel A: 10 mg Islatravir | Panel B: 2 mg Islatravir | Panel C: 30 mg Islatravir | Panel D: 1 mg Islatravir | Panel E: 0.5 mg Islatravir
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
hr*pmol/10^6 cells | 227 (33.3) | 46.9 (38.1) | 926 (47.7) | 35.9 (27.6) | 23.1 (83.0)

4. Secondary Outcome: Maximum Concentration (Cmax) of Islatravir Triphosphate in Peripheral Blood Mononuclear Cells
Description: Blood was collected to measure intracellular islatravir triphosphate concentration in peripheral blood mononuclear cells and determine Cmax.
Time Frame: as for outcome 3
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment, were compliant with study procedures, had Cmax of islatravir triphosphate in peripheral blood mononuclear cells data available, and were evaluable for the outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/10^6 cells
Arm/Group | Panel A: 10 mg Islatravir | Panel B: 2 mg Islatravir | Panel C: 30 mg Islatravir | Panel D: 1 mg Islatravir | Panel E: 0.5 mg Islatravir
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
pmol/10^6 cells | 2.81 (49.9) | 0.495 (62.9) | 8.9 (60.3) | 0.408 (49.3) | 0.263 (54.5)

5. Secondary Outcome: Concentration of Islatravir Triphosphate in Peripheral Blood Mononuclear Cells at 168 Hours Post-Dose (C168hr)
Description: Blood was collected to measure intracellular islatravir triphosphate concentration in peripheral blood mononuclear cells and determine C168hr.
Time Frame: 168 hours after islatravir administration
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment, were compliant with study procedures, had C168hr of islatravir triphosphate in peripheral blood mononuclear cells data available, and were evaluable for the outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/10^6 cells
Arm/Group | Panel A: 10 mg Islatravir | Panel B: 2 mg Islatravir | Panel C: 30 mg Islatravir | Panel D: 1 mg Islatravir | Panel E: 0.5 mg Islatravir
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
pmol/10^6 cells | 0.983 (26) | 0.188 (39.2) | 4.83 (85.9) | 0.164 (31.4) | 0.116 (85.6)

6. Secondary Outcome: Time to Maximum Concentration (Tmax) of Islatravir Triphosphate in Peripheral Blood Mononuclear Cells
Description: Blood was collected to measure intracellular islatravir triphosphate concentration in peripheral blood mononuclear cells and determine TMax.
Time Frame: as for outcome 3
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment, were compliant with study procedures, had Tmax of islatravir triphosphate in peripheral blood mononuclear cells data available, and were evaluable for the outcome measure.
Measure: Median (Full Range); unit: Hour
Arm/Group | Panel A: 10 mg Islatravir | Panel B: 2 mg Islatravir | Panel C: 30 mg Islatravir | Panel D: 1 mg Islatravir | Panel E: 0.5 mg Islatravir
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Hour | 12 [12 to 240] | 8 [4 to 144] | 24 [4 to 96] | 8 [4 to 24] | 12 [4 to 24]

7. Secondary Outcome: Apparent Terminal Half-Life (t1/2) of Islatravir Triphosphate in Peripheral Blood Mononuclear Cells
Description: Blood was collected to measure intracellular islatravir triphosphate concentration in peripheral blood mononuclear cells and determine apparent terminal t1/2.
Time Frame: as for outcome 3
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment, were compliant with study procedures, had apparent terminal t1/2 of islatravir triphosphate in peripheral blood mononuclear cells data available, and were evaluable for the outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Panel A: 10 mg Islatravir | Panel B: 2 mg Islatravir | Panel C: 30 mg Islatravir | Panel D: 1 mg Islatravir | Panel E: 0.5 mg Islatravir
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6
Hours | 128 (42.2) | 120 (14.7) | 78.5 (31.4) | 118 (16.1) | 95.3 (38.2)

8. Secondary Outcome: Area Under the Plasma Concentration-Time Curve of Islatravir From Time 0 to 168 Hours (AUC0-168hr)
Description: Blood was collected for the determination of AUC0-168hr of islatravir in plasma.
Time Frame: Predose and at 0.25, 0.5, 1, 2, 4, 8, 12, 24, 48, and 96 hours after islatravir administration. Value at 168 hours was extrapolated.
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment, were compliant with study procedures, had plasma AUC-168hr of islatravir data available, and were evaluable for the outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*nM
Arm/Group | Panel A: 10 mg Islatravir | Panel B: 2 mg Islatravir | Panel C: 30 mg Islatravir | Panel D: 1 mg Islatravir | Panel E: 0.5 mg Islatravir
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
hr*nM | 1020 (16.8) | 143 (39.6) | 3020 (24.6) | 88.3 (33.8) | 38.3 (25.8)

9. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Islatravir
Description: Blood was collected for the determination of Cmax of islatravir in plasma.
Time Frame: Predose and at 0.25, 0.5, 1, 2, 4, 8, 12, 24, 48, and 96 hours after islatravir administration
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment, were compliant with study procedures, had plasma Cmax of islatravir data available, and were evaluable for the outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Panel A: 10 mg Islatravir | Panel B: 2 mg Islatravir | Panel C: 30 mg Islatravir | Panel D: 1 mg Islatravir | Panel E: 0.5 mg Islatravir
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
nM | 235 (32.1) | 43.8 (51.2) | 678 (29.6) | 38.8 (31.3) | 20.3 (36.4)

10. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Islatravir
Description: Blood was collected for the determination of Tmax of islatravir in plasma.
Time Frame: Predose and at 0.25, 0.5, 1, 2, 4, 8, 12, 24, 48, and 96 hours after islatravir administration
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment, were compliant with study procedures, had plasma Tmax of islatravir data available, and were evaluable for the outcome measure.
Measure: Median (Full Range); unit: Hour
Arm/Group | Panel A: 10 mg Islatravir | Panel B: 2 mg Islatravir | Panel C: 30 mg Islatravir | Panel D: 1 mg Islatravir | Panel E: 0.5 mg Islatravir
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Hour | 1 [0.5 to 1] | 0.5 [0.5 to 1] | 0.75 [0.5 to 1] | 0.5 [0.5 to 1] | 0.5 [0.25 to 0.5]

11. Secondary Outcome: Apparent Terminal Half-Life (t1/2) of Islatravir in Plasma
Description: Blood was collected for the determination of apparent terminal t1/2 of islatravir in plasma.
Time Frame: Predose and at 0.25, 0.5, 1, 2, 4, 8, 12, 24, 48, and 96 hours after islatravir administration
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment, were compliant with study procedures, had apparent terminal t1/2 of islatravir in plasma data available, and were evaluable for the outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Panel A: 10 mg Islatravir | Panel B: 2 mg Islatravir | Panel C: 30 mg Islatravir | Panel D: 1 mg Islatravir | Panel E: 0.5 mg Islatravir
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Hours | 59.7 (15.4) | 47.4 (74.6) | 56.8 (11.2) | 10.4 (144) | 2.31 (16.7)

ADVERSE EVENTS:
Time Frame: Up to 21 days following administration of investigational drug
Description: All participants who received at least one dose of investigational drug
Arm/Group | Panel A: 10 mg Islatravir | Panel B: 2 mg Islatravir | Panel C: 30 mg Islatravir | Panel D: 1 mg Islatravir | Panel E: 0.5 mg Islatravir
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/6 | 5/6 | 6/6 | 5/6 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panel A: 10 mg Islatravir (N=6) | Panel B: 2 mg Islatravir (N=6) | Panel C: 30 mg Islatravir (N=6) | Panel D: 1 mg Islatravir (N=6) | Panel E: 0.5 mg Islatravir (N=6)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral mucosa erosion (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (6) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sensory disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Apathy (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-21): https://cdn.clinicaltrials.gov/large-docs/04/NCT02217904/Prot_SAP_000.pdf